CLINICAL TRIAL: NCT02211391
Title: The Effect of Nighttime Protein Intake on Overnight Lipolysis and Morning Fat Oxidation in Obese Men.
Brief Title: Nighttime Protein Intake on Overnight Lipolysis and Morning Fat Oxidation in Obese Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Assistant Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSC# 2014.13509
Record Dates: First submitted 2014-08-04; First posted 2014-08-07 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Obesity
Keywords: Nighttime Eating; Protein; Obesity; Lipolysis; Metabolism
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Casein Protein (Experimental): Casein protein (30g) will be consumed as the last food/caloric beverage and within 30 minute of sleep
  Interventions: Other: Casein Protein
- Non-caloric Placebo (Placebo Comparator): The non-caloric placebo beverage will will be consumed as the last food/caloric beverage and within 30 minute of sleep
  Interventions: Other: Non-caloric placebo

INTERVENTIONS:
Other: Casein Protein — The effect of casein protein consumed within 30 minutes of sleep on overnight lipolysis and next morning metabolism and appetite will be examined
  Arms: Casein Protein
Other: Non-caloric placebo — The effect of a non-caloric placebo consumed within 30 minutes of sleep on overnight lipolysis and next morning metabolism and appetite will be examined
  Arms: Non-caloric Placebo

SUMMARY:
Single macronutrients will be consumed before sleep by obese men. Overnight lipolysis will be measured with the microdialysis technique by measuring glycerol concentration and blood flow in abdominal adipose tissue. Morning fat oxidation will be measured with indirect calorimetry.

The investigators hypothesize that carbohydrate intake will blunt the overnight lipolysis rate compared to casein protein and a non-caloric placebo. The investigators also hypothesize that casein and placebo will not be significantly different from each other in terms of overnight lipolysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, sedentary overweight or obese (BMI ≥25 kg/m^2; body fat ≥ 25% ) men

Exclusion Criteria:

* Men that have been exercising for more than 2 days per week for more than 45 minutes per session (within the past 6 months), have uncontrolled hypertension (Blood Pressure (BP)>160/100 mmHg, diagnosed cardiovascular disease, stroke, diabetes, thyroid or kidney dysfunction, take cholesterol medication, or have any allergies to milk products will be excluded. Smokers will also be excluded.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Lipolysis | Change from day 1 to day 2 to day 3 of testing
  Measuring lipolysis using the microdialysis technique. Samples will be collected at various time intervals
  Vial 1: 30 minute; 2.0 uL/min flow rate
  Vial 2: 4 hours; 0.3 uL/min flow rate
  Vial 3: Overnight; 0.3 uL/min flow rate (before taking nighttime supplement)
  Vial 4: Morning sample #1; 2.0 uL/min flow rate (upon waking)
  Vial 5: Morning sample #2; 2.0 uL/min flow rate (arrive to lab)
  Blood flow will be measured using the Ethanol technique

SECONDARY OUTCOMES:
Resting Metabolic Rate (RMR) | Change from day 1 to day 2 to day 3
  RMR will be measured with indirect calorimetry using the ventilated hood technique

OTHER OUTCOMES:
Appetite | Change from Baseline to day 1, 2, and 3
  Appetite will be measured by visual analog scales
Blood hormones | Change from Baseline to day 1, 2, and 3
  Hormones related to appetite and metabolism will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Ormsbee, PhD, Principal Investigator — Florida State University
Locations (1):
- Institute of Sports Science and Medicine, Florida State University, Tallahassee, Florida, United States